CLINICAL TRIAL: NCT03319303
Title: Observational Study of the Effect of Tracheal Intubation and Tracheal Tube Position on Regional Lung Ventilation During General Anaesthesia
Brief Title: What Effect Does Intubation Have on Regional Lung Ventilation?
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: AN17/97842
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During any general anaesthetic which involves muscle relaxation artificial breathing is required. This is most commonly provided by pushing air under pressure (positive pressure ventilation) into the lungs via a tube in the airway (the tracheal tube). It has been observed for many years that with this form of breathing the distribution of gas within the lungs differs from that seen during 'natural' breathing: more of the gas goes to the upper parts of the lung than lower parts. This change in how the gas is distributed can lead to problems with how well oxygen is taken up by blood and carbon dioxide removed from the body. Previous work using mathematical modelling has found that the position of the tracheal tube might affect air distribution, but this has previously been difficult to study in 'real life', requiring the use of radioactive dyes and computerised tomography (CT). However a bedside test is now available which allows us to study these changes rapidly and non-invasively, using electrical impedance tomography (EIT). The EIT device is commercially available (PulmoVista®, Draeger UK) and is used in hospitals worldwide as a bedside monitor of lung ventilation.

This study aims to investigate the effect of tracheal intubation on regional ventilation of the lungs by comparing measurements before and after the patient is anaesthetised and intubated. The investgiators aim to show whether altered patterns of ventilation are caused by patients simply being asleep and ventilated, or whether these changes are due to the use of a tracheal tube itself. The exact effect of tube position will also be studied by measuring ventilation as the tube is deliberately advanced until it enters one of the lungs. This will give us information about the ideal position for a tube within the trachea to promote optimal ventilation patterns within the lungs

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to consent
2. undergoing a surgical procedure for which the anaesthetic technique includes muscle relaxation, intubation and ventilation for clinical care.

Exclusion Criteria:

1. Unwilling or unable to consent
2. co-existant respiratory disease associated with known abnormalities of ventilation/perfusion matching. This includes chronic obstructive pulmonary disease, asthma, or abnormalities of the chest wall or abdomen affecting ventilation e.g. morbid obesity
3. Requirement for double-lumen tracheal tube for clinical care
4. increased risk of regurgitation/aspiration e.g. pregnancy, symptomatic acid reflux, structural abnormalities of the gastro-intestinal tract (e.g. hiatus hernia)

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients attending for a surgical procedure are eligible and will be approached.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Manipulation of the tracheal tube and deliberate insertion into a right or left main bronchus | 20 mins
  General anaesthesia will then be induced, and when the participant is asleep a further set of measurements will be taken using the Electrical impedance tomography (EIT) belt whilst ventilation is maintained using the normal bag-mask ventilation technique used by anaesthetists in the first few minutes of the anaesthetic. Following this, the trachea will be intubated by the anaesthetist clinically responsible for the patient, and a further set of EIT measurements taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom